CLINICAL TRIAL: NCT06229652
Title: The Impact of Stress Management Interventions on Stress Perception, Coping Strategies, and Residual Symptoms in Depression: a Randomized Controlled Trial Investigating Psychological, Biological, Epigenetic, and Brain Correlates
Brief Title: Stress Management in Depressive Disorder: Resilience Training vs. Yoga: Biological, Epigenetic, and Brain Correlates
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Collaborators: University of Innsbruck (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Coping with Stress in MDD
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-01

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Stress management; Coping; Resilience; Yoga
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RASMUS Resilience Training (Experimental): RASMUS is a systematic, behavior-oriented group training in which the following methods are used: mindfulness exercises, exercises in self-compassion/guided meditations, knowledge transfer by means of a teaching talk/lecture, working out the topics in individual and small group work, group exercises, group discussion and exchange, train coping strategies: somatic, cognitive, and emotional levels, independent reflection on what has been learned, homework, weekly protocols, transfer to everyday life, questionnaires on resilience factors, mindfulness, and self-compassion for self-control, linking the course topics with one another.
  Interventions: Behavioral: RASMUS Resilience Training
- Body-oriented Yoga (Active Comparator): The body-oriented yoga classes following the Ashtanga style will run in parallel to the RAMUS resilience group (one-hour, once a week). The yoga instructor will support each participant in the form of verbal and hands-on assistance.
  Interventions: Other: Body-oriented Yoga

INTERVENTIONS:
Behavioral: RASMUS Resilience Training — RASMUS stands for "Resilience through mindfulness, self-compassion and self-care" and is a German-language 10-week group resilience program with one training unit per week. The main content of the RASMUS is based on seven resilience factors, i.e. acceptance, optimism, taking responsibility, solution orientation, future orientation, role clarity, and network orientation including the aspects of mindfulness, self-compassion, and self-care.
  RASMUS has been tested and certified according to the German Prevention Standard. The Central Prevention Test Center has awarded the seal of approval for the areas of exercise, nutrition, stress management/relaxation, and addictive substance consumption. Accordingly, this training program has been certified as a prevention course that is recognized by the German statutory health insurance companies. Furthermore, RASMUS can and is already offered as a (group) online course.
  Arms: RASMUS Resilience Training
Other: Body-oriented Yoga — Body-oriented Yoga following the Ashtanga style will be held by certified yoga teacher parallel to the experimental one hour per week 10 times.
  Each yoga session will start with the proper warming up of the whole body with some stretching exercises (20 min). The main part will last about 30 minutes and consist of dynamic and active yoga sequencing containing sun salutation with a mix of exercises. A relaxation phase with controlled breathing and meditation-elements will finish the class (10 min). Each exercise has different complexity levels of implementation and will be adapted to the performance abilities of each participant.
  Arms: Body-oriented Yoga

SUMMARY:
The aim of this clinical trial is to evaluate the effects of a Resilience and Stress Management Intervention Program (RASMUS) compared with yoga on stress perception, coping strategies, depressive symptoms, anxiety, resilience and quality of life in people diagnosed with major depressive disorder (MDD) in the short and long term.

In addition to psychological factors, biological parameters will be examined to define biomarkers involved in stress response. In the optional neuroimaging part, the effects of the planned interventions on the structure, metabolism and function of the brain will be investigated. The epigenetic part, which is also optional, will examine the effects of the planned interventions on the histone modifications.

DETAILED DESCRIPTION:
The aim of this clinical trial is to evaluate the effects of a Resilience and Stress Management Intervention Program (RASMUS) compared with yoga on stress perception, coping strategies, depressive symptoms, anxiety, resilience and quality of life in people diagnosed with major depressive disorder (MDD) in the short and long term.

In addition to psychological factors, biological parameters will be examined to define biomarkers involved in stress response. In the optional neuroimaging part, the effects of the planned interventions on the structure, metabolism and function of the brain will be investigated. The epigenetic part, which is also optional, will examine the effects of the planned interventions on the histone modifications. A total of 80 participants per study arm are planned for both the MRI and epigenetic studies (20 per gender and per type of intervention).

150 outpatients diagnosed with MDD will be randomly assigned to one of two groups: an experimental group receiving RASMUS training, and a control group receiving body-oriented yoga. Both interventions will take place in a group setting of 10-12 participants once a week for one hour over a period of 10 weeks. RASMUS aims to build, reflect on and strengthen stress management strategies and resilience through mindfulness, self-compassion and self-care. Through body-oriented yoga, participants learn through physical exercises to better control and manage their perception of stress.

The planned duration of the clinical trial is 4 years. Individual participation in the study will last approximately 8 months and include 4 study visits. The first visit will take place after enrolment. The second and third visits will take place after the fifth and final intervention. The fourth visit will be six months later.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MDD,
* Outpatient care for at least 3 months,
* Ongoing psychopharmacological treatment,
* Age between 18 and 65 years,
* Knowledge of written and spoken German,
* MADRS score ≤ 34 (moderate severity of symptoms),
* Written informed consent.

Exclusion Criteria:

* Other Axis I psychiatric disorder (organic mental disorders, psychoactive substance use [excl. caffeine and nicotine abuse], schizophrenia, bipolar disorder, neurotic disorders [excl. anxiety disorders], eating disorders, acute suicidality)
* Severe somatic illnesses,
* Pregnancy/breastfeeding,
* Undertaking regular yoga practice (more than once per week) over the past 3 months,
* Current use of psychotherapy.

Further exclusion criteria for the neuroimaging sub-study:

* History of neurological trauma or trauma to the central nervous system,
* MRI contraindications (claustrophobia, metallic, electrical, magnetic or mechanically driven implants, tattoos on the head or neck or other clinically relevant contraindications)
* Positive drug urine test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Total Change Scores on the Stress Processing Questionnaire (SVF-ak) among Study Completers | 0 weeks (baseline), 10 weeks (post treatment) (post1) and 6-months follow-up (post2)
  Stress perception and stress processing modes in the sense of state characteristics will be assessed with the Stress Processing Questionnaire (SVF-ak) (Janke & Erdmann, 1997; Janke et al., 1985; Kühn, 1986). The SVF-ak retrospectively asks about the stress processing methods used during a previous stress phase/period. The short version of this instrument which will be used in this study consists of 42 questions for the assessment of the extent to which the 19 processing strategies of the SVF - supplemented by the subtest helplessness - were used in certain stressful situations. Subjects indicate on a 4-point scale ranging from 0 (in no case) to 3 (for sure/ with certainty), how often the thought formulated in the item "went through their mind in the previous situation".
Total Change Scores on the Perceived Stress Scale (PSS-10) among Study Completers | 0 weeks (baseline), 10 weeks (post treatment) (post1) and 6-months follow-up (post2)
  The German version of the Perceived Stress Scale (PSS-10) by Klein et al. (2016) will be used to measure excessive demands and the perception of stress. Subjects indicate on a 5-point Likert scale ranging from null (never) to four (very often) the extent to which situations in their own lives were unpredictable, uncontrollable, and overwhelming in the past month.

SECONDARY OUTCOMES:
Total Change Scores on the State-Trait-Anxiety Inventory (STAI) among Study Completers | 0 weeks (baseline), week 5 (mid), 10 weeks (post treatment) (post1) and 6-months follow-up (post2)
  Assessment of present and long-lasting anxiety levels will be carried out with the State-Trait-Anxiety Inventory (STAI) (Spielberger et al., 1970, German version by Laux et al., 1981). This is a widely used 40-items multiple-choice questionnaire assessing two dimensions of anxiety: anxiety as a trait (STAI-T), and anxiety as a transient emotional state (STAI-S). The STAI comprises 20 anxiety-related items rated on a 4-point Likert-scale ranging from 1 (not at all) to 4 (totally). Total scores range from 20 to 80 with higher scores indicating higher anxiety. Both state and trait anxiety will be assessed at baseline. At the other time points (mid, post1, post2) only state anxiety will be assessed.
Total Change Scores on the Resilience Scale for Adults (RSA) among Study Completers | 0 weeks (baseline), 10 weeks (post treatment) (post1) and 6-months follow-up (post2)
  Resilience will be evaluated using the Resilience Scale for Adults (RSA; Friborg, 2003; German version by Kaiser et al., 2019). This scale consists of 33 items rated on a 7-point intensity response scale and is used to measure both intra- and interpersonal protective factors. These protective factors promote adaptation to adversity and are examined in the following areas: self-perception, future planning, social competence, structural style, family cohesion, and social resources. Mean scores within each subscale are calculated or the total score.
Total Change Scores on the WHO Quality of Life - Brief Version (WHOQOL-BREF) among Study Completers | 0 weeks (baseline), 10 weeks (post treatment) (post1) and 6-months follow-up (post2)
  Subjectively perceived quality of life will be assessed with the WHO Quality of Life - Brief Version quality of life measure (WHOQOL-BREF; Skevington et al., 2004). This is a 26-item self-report questionnaire to assess quality of life over the past two weeks in four domains: physical, psychological, social, and environmental. The items are rated on a five-point Likert scale from 1 (absent) to 5 (severe). The total scale is used in this study with higher scores indicating better quality of life.
Total Change Scores on the Beck Depression Inventory-II (BDI-II) among Study Completers | 0 weeks (baseline), week 5 (mid), 10 weeks (post treatment) (post1) and 6-months follow-up (post2)
  The primary outcome - severity of depressive symptoms will be evaluated by means of the Beck Depression Inventory-II (BDI-II) (Beck et al., 1996; German translation by Kühner et al., 2007). The BDI-II is a 21-item self-report questionnaire to assess the severity of depression in the past two weeks. Each question has a set of four possible responses, ranging in intensity and resulting in a maximum total score of 63. Higher total scores indicate more severe depressive symptoms. BDI scores between 0 and 13 indicate absent to minimal depressive symptoms, from 14 to 19 mild symptoms, from 20 to 28 moderate symptoms, and from 29 to 63 severe depressive symptoms.
Total Change Scores on the Montgomery-Asberg Depression Rating Scale (MADRS) among Study Completers | 0 weeks (baseline), 10 weeks (post treatment) (post1) and 6-months follow-up (post2)
  The severity of (residual) depressive symptoms will be evaluated using the MADRS. This observer-rated interview consists of 10 items (apparent sadness, reported sadness, internal tension, decreased sleep, decreased appetite, difficulty concentrating, fatigue, inability to feel, as well as pessimistic and suicidal thoughts), with each item scoring from 0 to 6. The total score ranges from 0 to 60 with higher scores reflecting a higher severity of symptoms. MADRS score ranging from 0 to 6 indicates absent to minimal depressive symptoms, from 7 to 19 mild depression, from 20 to 34 moderate depression, score of 35 and greater indicates severe symptoms and score of 60 indicates very severe depression.
Alcohol/ tobacco consumption | 0 weeks (baseline), 10 weeks (post treatment) (post1) and 6-months follow-up (post2)
  Alcohol/ tobacco consumption will be assessed using the Tobacco and Alcohol Questionnaire (Sánchez-Gutiérrez et al., 2023)

OTHER OUTCOMES:
Total Change Scores on the Positive and Negative Affect Schedule (PANAS) | 0 weeks (baseline), week 5 (mid), 10 weeks (post treatment) (post1) and 6-months follow-up (post2)
  The degree of engagement, immediate response, and changes in affective state will be monitored before and after the first, fifth, and tenth training unit using the Positive and Negative Affect Schedule (PANAS) (German version by Breyer & Bluemke, 2016). This questionnaire consists of 20 adjectives that describe various feelings and emotions and are rated on a five-point scale from "not at all" to "very much". Ten adjectives each capture the dimensions of positive and negative affect. The result is the sum of the values.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Hofer, Dr., Study Director — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria